CLINICAL TRIAL: NCT04265196
Title: Group Therapy for Fibromyalgia: RCT Testing the Effectiveness of Mindfulness -Based Therapy Versus Cognitive-behavioral Therapy
Brief Title: Group Therapy for Fibromyalgia:the Effectiveness of Mindfulness -Based VS Cognitive-behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bar-Ilan University, Israel (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Principal Investigator, Danny Horesh, Senior lecturer and head of the Trauma and Stress Research Lab at Bar-Ilan University's Department of Psychology., Bar-Ilan University, Israel
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 10112019
Record Dates: First submitted 2020-02-02; First posted 2020-02-11 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Fibromyalgia; PTSD; Depression; Stress; Sleep Disturbance
MeSH Terms: conditions — Fibromyalgia; Stress Disorders, Post-Traumatic; Depression; Parasomnias

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be assigned to the different treatment groups randomly and without receiving information about the different treatment options included in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cognitive behavioral group therapy (Experimental): A Cognitive Behavioral Therapy intervention is based on a unique protocol built in the light of previous research in the field and includes a 10-week treatment focused on coping with pain and stress.
  Interventions: Other: cognitive behavioral group therapy
- Mindfulness-based group therapy (Experimental): A mindfulness-based group therapy intervention was built inspired by a mindfulness protocol that is effective in treating pain, and includes adjustments to the physical distress of fibromyalgia patients as well as an emphasis on coping with stress and pain.
  Interventions: Other: Mindfulness-based group therapy
- control group (No Intervention): A control group will wait for 3 months, during which the subjects will complete the questionnaires and only after the end of the period will they participate in the treatment so that it will serve as a control group without intervention.

INTERVENTIONS:
Other: cognitive behavioral group therapy — A unique protocol that includes cognitive-behavioral psychological therapy with emphasis on coping with pain
  Arms: cognitive behavioral group therapy
Other: Mindfulness-based group therapy — Unique protocol that includes mindfulness-based psychological therapy with emphasis on coping with pain
  Arms: Mindfulness-based group therapy

SUMMARY:
This study was conducted as part of a collaboration between the Maccabi Health Fund and Bar Ilan University. Fibromyalgia is a chronic pain disorder, highly co-morbid with depression, stress, and anxiety. the investigators aim to examine the effect of group cognitive-behavioral therapy (CBT) and mindfulness-based intervention (MBI) among fibromyalgia patients. the investigators will also examine which intervention fits which patient, according to one's individual characteristics, in hope that this would enable Maccabi to offer personalized treatment. Furthermore, the investigators wish to identify the underlying cognitive and psychopathological mechanisms (measured during treatment) by which each intervention works.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic pain disorder, highly co-morbid with depression, stress, and anxiety. the investigators aim to examine the effect of group cognitive-behavioral therapy (CBT) and mindfulness-based intervention (MBI) among fibromyalgia patients. the investigators will also examine which intervention fits which patient, according to one's individual characteristics, in hope that this would enable Maccabi to offer personalized treatment. Furthermore, the investigators wish to identify the underlying cognitive and psychopathological mechanisms (measured during treatment) by which each intervention works.

First, the investigators expect that CBT and MBI will lead to greater improvement in physical, psychological, and behavioral measures among fibromyalgia patients compared to waitlist controls. Second, the investigators expect that MBI and CBT will have a differential effect, so that some outcome variables will show greater improvement following one intervention, but not the other. Furthermore, factors such as age, illness duration, symptom severity, and initial psychopathology levels will affect one's level of improvement following these interventions. Finally, the investigators expect to identify differential mechanisms driving each intervention. The study is a randomized controlled trial (RCT), including 90 fibromyalgia patients, randomly assigned to 3 conditions: (1) Group CBT (n=30), (2) MBI (n=30), (3) Waitlist control group, subsequently assigned to treatment (n=30). Participants will complete selfreport questionnaires tapping psychological (depression, stress), cognitive (observing negative experiences "from afar", cognitive flexibility towards pain) and physical (pain, body awareness) aspects, at 4 assessments: pre-/during/post- treatment, and 3 months after treatment.

To date, no RCT comparing CBT and MBI for fibromyalgia was conducted. Comparing them would be highly important, as they are the two most notable psychological interventions for chronic pain conditions. This study would enable Maccabi to offer improved psychological services for fibromyalgia. Furthermore, group therapy may serve as an effective treatment meeting both Maccabi's needs (a short, economic intervention) and patients' needs (a condition-specific treatment, offering group support and stigma reduction).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with fibromyalgia
* Hebrew speakers

Exclusion Criteria:

* Patients who are actively suicidal
* Patients who suffering from psychotic status
* Patients who are chronically use addictive substances,
* Patients who had unusual cognitive or physical disability that would prevent them from participating in mindfulness exercises

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
The Fibromyalgia Impact Questionnaire Revised (FIQR) | change through study completion, an average of 6 month
  Self-report questionnaire, which includes 21 items and assesses symptoms and functioning of fibromyalgia patients, taking into account the frequency of symptoms, their intensity, and the degree of impairment of patient function
Perceived Stress Scale (PSS) | change through study completion, an average of 6 month
  A 10-item questionnaire measuring the level at which events occurred in the individual's life in the past month is perceived as unpredictable, uncontrollable and overwhelming. A higher score indicates a higher level of perceived stress.
The Patient Health Questionnaire-9 (PHQ-9) | change through study completion, an average of 6 month
  A self-reported 9-item questionnaire to measure symptoms of major depression. The items relate to the key aspects of DSM, including thoughts of death, loss of appetite, sadness and mental pain, and negative cognitions.
Pain (VAS) | change through study completion, an average of 6 month
  Self-report questionnaire designed to measure pain intensity and unpleasantness caused by pain. This questionnaire is widely used in pain clinics. It includes one item that can be graded on a continuous scale that ranges from 0 (no pain) to 10 (the worst pain that can be).
Sleep Quality (Pittsburgh Sleep Quality Index) | change through study completion, an average of 6 month
  A questionnaire developed to measure sleep quality and sleep disorder. The questionnaire includes 19 items measuring seven components of sleep (sleep quality, sleep onset, sleep duration, sleep efficiency, sleep disturbance, sleep medication use, and daily functioning impairment) over the past four weeks.

SECONDARY OUTCOMES:
Mindfulness (Five Fact Mindfulness Questionnaire) | change through study completion, an average of 6 month
  The questionnaire includes 5 scales, which relate to various mindfulness factors - observing / paying attention to internal and external stimuli , the ability to verbally describe or label stimuli, behavior, non-judgmental and non-reactivity
Psychological Inflexibility in Pain (PIPS) | change through study completion, an average of 6 month
  A questionnaire designed to assess the extent to which a person is trying to control and struggle with physical pain, as opposed to trying and accepting it, and "making friends" with him. The questionnaire includes 12 items.
Body Vigilance (BVS) | change through study completion, an average of 6 month
  Self-report questionnaire designed to examine attention regarding normal physical processes, periodic susceptibility / rhythm sensitivity, and ability to predict physical responses. Each item in the questionnaire is rated on a 7-rank Likert scale (1 = not at all true, 7 = very true), with a higher score representing a higher body awareness.
Meta-cognition (MCQ-30) | change through study completion, an average of 6 month
  A self-report questionnaire designed to test metacognitive ability, with an emphasis on beliefs, judgment, and regulation.
Difficulties in emotion regulation (DERS) | change through study completion, an average of 6 month
  Self-report questionnaire designed to test difficulties in the emotional regulation process. The questionnaire contains 36 items that relate to awareness of emotions and emotional reactions
Pain Catastrophizing (PCS) | change through study completion, an average of 6 month
  A questionnaire examining the tendency to intensify the threat and sense of helplessness arising from pain, and the inability to prevent it
Trauma Exposure (The Life Events Checklist) | Pre-treatment
  An index that examines exposure to traumatic life events. Exposure is rated at various levels (direct, indirect, experience)
Self- Compassion (SCS) | change through study completion, an average of 6 month
  Self-report questionnaire that examines the participant's compassionate ability. The questionnaire refers to 3 components of compassion - Self-Kindness, Common Humanity and Mindfulness
Distress tolerance | change through study completion, an average of 6 month
  Self-report questionnaire covering four different categories: perceived ability to bear emotional distress, subjective assessment of distress, attentiveness to negative emotions, and regulation efforts to reduce distress.
  A combination of categories allows for an overall measure of distress resistance
Alexithymia | change through study completion, an average of 6 month
  Self-Reporting Questionnaire Examining three subscales: (1) difficulty identifying feelings and distinguishing between feelings and bodily sensations in emotional activation, (2) difficulty in the verbal expression of emotions, and (3) externally oriented thinking.

CONTACTS AND LOCATIONS:
Overall Officials: Danny Horesh, Phd, Principal Investigator — Bar Ilan University
Locations (1):
- Bar Ilan University, Ramat Gan, Israel